CLINICAL TRIAL: NCT03095521
Title: A Prospective, Multi-center, Open, Randomized Clinical Study in Parallel Groups, for the Comparative Evaluation of Efficacy and Safety of Angal, Lozenges [Menthol], 1 mg + 5 mg (Sandoz d.d., Slovenia), and ANTI-ANGIN® FORMULA, Lozenges, 0,2 mg + 2 mg + 50 mg (LLC "Valeant", Russia) in Treatment of Patients With Uncomplicated Acute Infectious and Inflammatory Diseases of the Pharynx, Accompanied by a Sore Throat.
Brief Title: A Local Clinical Study for the Comparative Evaluation of Efficacy and Safety of Angal, Lozenges [Menthol] and ANTI-ANGIN® FORMULA, Lozenges, in Treatment of Patients With a Sore Throat
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TE_004_ANG_LOZ
Record Dates: First submitted 2017-03-21; First posted 2017-03-29 (Actual); Results first posted 2019-03-22 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2018-12

CONDITIONS: Sore Throat
Keywords: Angal; ANTI-ANGIN® FORMULA; sore throat; no less therapeutic efficacy
MeSH Terms: conditions — Pharyngitis | interventions — Menthol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Angal, lozenges, per 1 lozenge, with an interval 2 hours or more, 6-10 lozenges per day, for a maximum 4 days or until full illness resolution, if this will happen earlier than 4th day of treatment.
  Interventions: Drug: Angal, lozenges [menthol],
- Arm B (Active Comparator): ANTIANGIN ® FORMULA, 1 lozenge, with an interval 2 hours or more, up to 6 lozenges per day, for a maximum 5 days or until full illness resolution, if this will happen earlier than 5th day of treatment.
  Interventions: Drug: ANTI-ANGIN® FORMULA

INTERVENTIONS:
Drug: Angal, lozenges [menthol], — Angal, administered per 1 lozenge, with an interval 2 hours or more, 6-10 lozenges per day, for a maximum 4 days or until full illness resolution.
  Arms: Arm A
Drug: ANTI-ANGIN® FORMULA — 0,2 mg + 2 mg + 50 mg (LLC "Valeant", Russia). Administered per 1 lozenge, with an interval 2 hours or more, up to 6 lozenges per day, for a maximum 5 days or until full illness resolution.
  Arms: Arm B

SUMMARY:
The purpose of this study was to evaluate no less therapeutic efficacy and safety of the Angal, lozenges [Menthol], 1 mg + 5 mg (Sandoz dd, Slovenia) compared to ANTI-ANGIN® FORMULA, lozenges, 0,2 mg + 2 mg + 50 mg (LLC "Valeant", Russia) in treatment of patients with uncomplicated acute infectious and inflammatory diseases of the pharynx, accompanied by a sore throat.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent for participation in this clinical study; 18 to 45 years old inclusive, male and female;
* Diagnosed uncomplicated acute infectious and inflammatory diseases of the pharynx, accompanied by a sore throat;
* Onset of first symptoms of the uncomplicated acute infectious and inflammatory diseases of the pharynx (pharyngitis and/or tonsillitis) less than 48 hours prior to inclusion into the study;
* Baseline TSS score (Tonsillopharyngitis Severity Score) ≥ 5 (total score);

Exclusion Criteria:

* Use of analgesics within <12 hours prior to the study start or/and inability to cancel them during the study;
* Use of antibiotics within <48 hours prior to the study start or/and inability to cancel them during the study;
* Use of local therapy (sprays, rinses, lozenges) to pharynx within <12 hours before study start or/and inability to cancel them, besides study medications.
* Use systemic or inhaled corticosteroids within ≤1 months prior to the study start and planned therapy of them during the study (besides skin means).
* Presence of symptoms of primary bacterial pharyngitis or secondary bacterial infection (including fever over 37,5 ° C, the presence of purulent raids in the throat, severe intoxication, leukocytosis, neutrophilia, shift leukocyte left (increasing the percentage of neutrophils sticks appearance younger forms of neutrophils), increased ESR 30 mm/hr);

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2017-05-07 (Actual); Study Completion 2017-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz, Study Director — Sandoz
Locations (4):
- Russia (4):
  - Sandoz Investigational Site, Arkhangelsk
  - Sandoz Investigational Site, Moscow
  - Sandoz Investigational Site, Saint Petersburg
  - Sandoz Investigational Site, Stavropol

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial included a screening period, up to 5 days active treatment, and follow-up visit. The patients had to visit the trial site up to 3 times.
Pre-assignment Details: 228 patients in total were included
Groups:
- ANGAL: Patients received Angal, lozenges, per 1 lozenge, with an interval 2 hours or more, 6-10 lozenges per day, for a maximum 4 days or until full illness resolution, if happened earlier than 4th day of treatment.
- ANTIANGIN: Patients received ANTIANGIN ® FORMULA, 1 lozenge, with an interval 2 hours or more, up to 6 lozenges per day, for a maximum 5 days or until full illness resolution, if happened earlier than 5th day of treatment.
Period: Overall Study
Arm/Group | ANGAL | ANTIANGIN
Started (231 screened, 3 excluded (breach in incl. criteria (2) and no hematology analyses (1)) | 115 | 113
Intent to Treat Population ITT | 115 | 113
Per Protocol Population PP | 113 | 107
Safety Population | 115 | 113
Completed | 115 | 111
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ANGAL | ANTIANGIN | Total
Number analyzed (Participants) | 115 | 113 | 228
Age, Continuous [Mean (Full Range); unit: years] — Population: ITT
  years | 30.44 [18 to 51] | 30.02 [18 to 45] | 30.23 [18 to 51]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: ITT
  Participants
    Female | 73 | 67 | 140
    Male | 42 | 46 | 88
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 115 | 113 | 228
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Without Sore Throat According to TSS Score
Description: TSS (Tonsillopharyngitis Severity Score) is a questionnaire for evaluation of the five following symptoms severity: pharyngalgia, difficulty in swallowing, salivation, hyperemia of pharyngeal mucosa, and body temperature increase according to a 4-point scale:
  0 : no symptoms
  1. : insignificant symptom
  2. : moderate symptom
  3. : significant symptom fever
  0 pts : <37.5 °С;
  1. pts : 37.5 to <38.5 °С;
  2. pts : 38.5 to <39.5 °С;
  3. pts : ≥ 39.5 °С. TSS total ranges are 0-15.
Time Frame: 4 days
Population: ITT, only patients with measurements were included (115 for Angal, and 112 for Antiangin)
Measure: Number; unit: percentage of participants
Arm/Group | ANGAL | ANTIANGIN
Number analyzed (Participants) | 115 | 112
percentage of participants
  sore throat TSS score 0 | 84.35 | 73.21
  sore throat TSS score 1 | 13.91 | 17.86
  sore throat TSS score 2 | 1.74 | 8.93
  sore throat TSS score 3 | 0 | 0
Statistical Analysis 1: Comparison: ANGAL vs ANTIANGIN; Arm Angal, Arm Antiangin; Test type: Non-Inferiority — two-sided 95% CIs estimation used to confirm non-inferior efficacy in primary endpoint. A non-inferiority conclusion was made relating to the primary parameter only; p = 0.028, Fisher Exact

2. Secondary Outcome: 50% Reduction Tss SCORE
Description: Frequency of 50 % or more total score reduction by the TSS questionnaire completed by the Investigator relative to baseline in both Angal and ANTI-ANGIN FORMULA arms at visit 2
Time Frame: day 4
Population: PP set was considered for the analysis, however only the number of patients with complete data at visit 2 were considered for the analysis
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ANGAL | ANTIANGIN
Number analyzed (Participants) | 110 | 105
percentage of participants | 97.35 [92.44 to 99.45] | 98.13 [93.41 to 99.77]

3. Secondary Outcome: Change From Baseline in TSS Total Score
Description: Change from baseline in TSS total score. A negative change from baseline means an improvement.TSS (Tonsillopharyngitis Severity Score) is a questionnaire for evaluation of the five following symptoms severity: pharyngalgia, difficulty in swallowing, salivation, hyperemia of pharyngeal mucosa, and body temperature increase according to a 4-point scale:
  0 : no symptoms
  1. : insignificant symptom
  2. : moderate symptom
  3. : significant symptom fever
  0 pts : <37.5 °С;
  1. pts : 37.5 to <38.5 °С;
  2. pts : 38.5 to <39.5 °С;
  3. pts : ≥ 39.5 °С. TSS total ranges are 0-15.
Time Frame: baseline and day 4
Population: PP
Measure: Mean (Full Range); unit: unit on a scale
Arm/Group | ANGAL | ANTIANGIN
Number analyzed (Participants) | 113 | 107
unit on a scale
  baseline | 6.88 [6.63 to 7.14] | 7.03 [6.75 to 7.30]
  day 4 | 0.45 [0.31 to 0.60] | 0.83 [0.57 to 1.08]

4. Secondary Outcome: Days to Recovery, Defined by the Patient's Diary (Subjective Evaluation by the Patient)
Description: only patients for which outcomes were available were included , 111 out of 113 for Angal and 102 out of 107 for Antiangin, per protocol set
Time Frame: 5 days
Population: PP
Measure: Mean (Standard Error); unit: days
Arm/Group | ANGAL | ANTIANGIN
Number analyzed (Participants) | 111 | 102
days | 3.75 (0.049) | 3.93 (0.059)
Statistical Analysis 1: Comparison: ANGAL; Test type: Superiority; p = 0.482, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Number of Participants Who Fully Recovered up to Day 5
Description: Number of participants who fully recovered up to day 5 (the outcome of a disease according to the objective evaluation by the Investigator, the total score according to the TSS questionnaire ≤ 2)
Time Frame: 4 days for Angal, 5 days for AntiAngin
Population: PP
Measure: Number; unit: participants
Arm/Group | ANGAL | ANTIANGIN
Number analyzed (Participants) | 113 | 107
participants | 102 | 104

6. Secondary Outcome: Change From Baseline in Sore Throat Intensity by 100 mm in Visual Analogue Scale Filled in by the Patient (VAS) .
Description: The VAS is a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." The VAS ranges from 0 to 100. A decrease from baseline in the VAS score to reflect pain intensity indicates a decrease in pain intensity.
Time Frame: baseline, day 4
Population: PP, participants with measure
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | ANGAL | ANTIANGIN
Number analyzed (Participants) | 113 | 107
millimeters
  Baseline | 66.38 (17.60) | 66.99 (18.03)
  day 4: number analyzed (Participants) | 113 | 106
  day 4 | 2.35 (7.96) | 4.67 (10.67)
Statistical Analysis 1: Comparison: ANGAL vs ANTIANGIN; change from baseline, 2 groups; Test type: Superiority; p = 0.072, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 5 days
Arm/Group | ANGAL | ANTIANGIN
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/113
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/113
Other Adverse Events (participants affected / at risk) | 6/115 | 12/113
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANGAL (N=115) | ANTIANGIN (N=113)
Sinus Tachicardia (Cardiac disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 1 (2)
hypoesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (2)
pyrexia (General disorders) | 0 (0) | 1 (1)
ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
red blood cell analysis abnormal (Investigations) | 1 (1) | 0 (0)
dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
pharyngeal hypoesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However Novartis does not prohibit any inversdtigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-09-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT03095521/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT03095521/SAP_001.pdf